CLINICAL TRIAL: NCT06609915
Title: SuprAglottic superImposed High Frequency Jet Ventilation veRsus High-flow nAsal oxYgen in Tubeless Laryngotracheal Surgery (AIRWAY): a Prospective Randomised Controlled Trial
Brief Title: SuprAglottic Jet Ventilation vs High-flow Nasal Oxygen in Tubeless Laryngotracheal Surgery
Acronym: AIRWAY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AIRWAY
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Airway Managment; Laryngotracheal Surgery

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Supraglottic, superimposed high frequency jet ventilation using the Monsoon 4 (Thora Tech GmbH, Giessen, Germany) with initial 1.0 FiO2 reduced to 0.3 during laser surgery
  Interventions: Device: supraglottic superimposed high frequency jet ventilation ventilation using the Monsoon 4 (Thora Tech GmbH, Giessen, Germany)
- Control group (Active Comparator): high-flow oxygen (up to 70 L/min FiO2 1.0) via nasal cannula with the Optiflow (Fisher & Paykel Healthcare, Auckland, New Zealand) with initial 1.0 FiO2 reduced to 0.3 during laser surgery
  Interventions: Device: High-flow nasal supplemental oxygen via nasal cannula with the Optiflow (Fisher & Paykel, Auckland, New Zealand)

INTERVENTIONS:
Device: supraglottic superimposed high frequency jet ventilation ventilation using the Monsoon 4 (Thora Tech GmbH, Giessen, Germany) — supraglottic superimposed high frequency jet ventilation ventilation using the Monsoon 4 (Thora Tech GmbH, Giessen, Germany). Initially FiO2 at 1.0, reduced to 0.3 during laser interventions. Frequency and pressure set according to the local standards
  Arms: Intervention group
Device: High-flow nasal supplemental oxygen via nasal cannula with the Optiflow (Fisher & Paykel, Auckland, New Zealand) — up to 70 L/min FiO2 1.0 high flow oxygen via nasal cannula with the Optiflow (Fisher & Paykel, Auckland, New Zealand) initially. Reduced FiO2 to 0.3 during laser intervention.
  Arms: Control group

SUMMARY:
This study aims to investigate two oxygenation methods (high flow nasal oxygen and supraglottic, superimposed high-frequency jet ventilation) for tubeless laryngotracheal surgeries concerning their safety and efficiency.

DETAILED DESCRIPTION:
Eligible adult patients will be prepared for intubation according to the local SOPs of the anesthesia departments. Mandatory monitoring will consist of: SpO2, HR, NIBP, tcCO2, EEG, TOF and EIT.

Induction of anesthesia: Patients will be preoxygenated before induction of anesthesia for at least one minute through face-mask with FiO2 1.0 until etO2 reaches 0.9. The induction of anesthesia will be performed using a combination of sedative/hypnotic drugs, opioids and muscle relaxant.

The following medications will be mandatory as per protocol:

* A neuromuscular blocking agent (NMBA): Rocuronium 0.5-1 mg/kg
* Propofol 1-3 mg/kg
* Opioid: Fentanyl 1-3mcg/kg, Remifentanyl 1-3mcg/kg

After induction of anesthesia and the administration of a NMBA, bag-mask ventilation with FiO2 1.0 will be performed for at least 60 seconds or until the muscle relaxant is working. Full neuromuscular blockade will be assessed by train-of-four (TOF) monitoring. Anaesthesia will be given total intravenously with Propofol and Remifentanil under EEG guidance. Tracheal tube will be placed recruitment manoeuver (RM) will be performed before surgical disinfection. The RM consists of recruitment pressure of 30 cmH2O during 30 seconds. PEEP level will be set at 10cmH20.

Thereafter placement of the surgical laryngoscope will be performed by the ENT-surgeon and the oxygenation device according to randomization will be installed. The patient will be extubated and the intervention start.

Jet ventilation Group (intervention-group): Patients will receive supraglottic superimposed high frequency jet ventilation using the Monsoon 4 (Thora Tech GmbH, Giessen, Germany), that will be directly attached to the operative suspension laryngoscope with a Luer-lock. Before use, pressure safety limits of the device will be tested. Initially FiO2 will remain at 1.0, FiO2 will be reduced to 0.3 during laser interventions. Frequency and pressure will be set according to the local standards.

High-Flow Oxygen Group (control-group): Patients will receive high-flow oxygen (up to 70 L/min FiO2 1.0) via nasal cannula with the Optiflow (Fisher & Paykel Healthcare, Auckland, New Zealand). FiO2 will remain at 1.0, FiO2 will be reduced to 0.3 during laser interventions.

If the measured SpO2 falls below 80%, or if the measured tcCO2 rises above 70mmHg, surgical procedures will be interrupted. Additionally, if deemed necessary, rescue strategies will be performed at the discretion of the attending anesthesiologist, even if the predefined thresholds are not crossed. Rescue oxygenation or decarboxylation will be provided, this may include increasing the FiO2 to 100% or performing tracheal tube placement by the surgeon, determined by the anaesthesiologist in charge. If this change in airway strategy remains unsuccessful, the local difficult airway algorithm will be followed according to the SOP.

If the rescue airway management was successful and respiratory parameters return to baseline levels, the initial airway device according to randomisation will be reapplied. A permanent switch of airway strategy leads to study termination.

EIT will be measured using PulmoVista® 500 by Dräger, Lübeck, Germany, to visualize possible atelectasis formation and its progression over time. EIT is a non-invasive, radiation-free technique for the assessment of spatial and temporal ventilation distribution based on the changes in electrical properties of the tissue during the respiratory cycle. EIT measurements will be performed using a commercially available setup (PulmoVista 500, Draeger, Germany). A loose-fitting belt with 16 evenly spaced electrodes will be placed around the participant's chest in thoracic median plane. Small electrical currents are injected through adjacent electrodes in a rotating mode. Resulting potential differences are measured, and impedance distribution sampled at 30 Hz will be calculated by an automated linearized newton-raphson reconstruction algorithm. The device is suitable for assessment of jet ventilation and high flow.

Thoracic electrical impedance tomography measurements (each measurement will last 1 min) will be performed at the following time points: before induction of the anaesthesia; before the surgical procedure when the induction is terminated and recruitment manoeuvers have been performed; after the termination of the surgical procedure; before transport to the Post anaesthesia Care Unit (PACU); before the discharge from the PACU after 2 hours of monitoring. Relative change in poorly ventilated lung. regions (silent spaces) and end-expiratory lung impedance (EELI) and measures of ventilation inhomogeneity such as the global inhomogeneity index will be calculated as described previously, using customised code (Matlab R2021a, The MathWorks, Nattick, Massachusetts, USA).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients aged ≥18 years
* Patients requiring elective tubeless laryngotracheal surgery

Exclusion Criteria:

* Patients <18 years
* High risk of aspiration which concludes the consideration of using a tube in order to prevent aspiration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall number of cases without interruptions | 2 hours
  Number of cases using SSHFJV vs HFNO without interruption of the surgical procedure for rescue, during tubeless laryngo-tracheal surgery from placement of the laryngoscope to end of surgery.

SECONDARY OUTCOMES:
Time until desaturation | 2 hours
  Time until desaturation starting with laser surgery
Reason for change of airway strategy | 5 minutes
  Reason for change of airway strategy given by the attending
Duration of interruptions | 15 minutes
  Duration of surgical interruptions to permit rescue
Number of interruptions | 5 minutes
  Number of surgical interruptions to permit rescue
Overall anesthesia time | 3 hours
  Overall anesthesia time
Duration of desaturation | 5 minutes
  Duration of desaturation (SpO2 <80%)
Overall surgery time | 2 hours
  Overall surgery time
Duration of hypercapnia | 5 minutes
  Duration of hypercapnia (>70mmHg)
Value of oxygen level | 5 minutes
  Value of lowest recorded SpO2 in %
Value of carbon dioxide level | 5 minutes
  Value of highest recorded tcCO2 in mmHg
Respiratory complications | 24 hours
  Number of occurrences of respiratory complications before PACU-discharge and within 24 hours postoperatively, such as airway injury, cardiopulmonary resuscitation, bleeding, aspiration of gastric contents, post-extubation stridor, laryngospasm, bronchospasm, need for High Flow Nasal Oxygen (if not preoperatively on oxygen), need for low flow nasal oxygen (if not preoperatively on oxygen) or need for re-intubation will be recorded. Respiratory complications are defined as the need for re-intubation after being extubated, persistent stridor (even if oxygen is not required), respiratory failure, the occurrence of pneumothorax or the need for any additional diagnostic examination following respiratory problems (i.e., bronchoscopy, radiology).
End-expiratory lung impedance (EELI) after the end of induction before the surgical procedure. | 1 hour
  End-expiratory lung impedance (EELI) detected by using electrical impedance tomography (EIT) after the end of induction before the surgical procedure.
End-expiratory lung impedance (EELI) at the end of the surgical procedure. | 3 hours
  End-expiratory lung impedance (EELI) detected by using electrical impedance tomography (EIT) at the end of the surgical procedure.
End-expiratory lung impedance (EELI) after the end of anaesthesia. | 3 hours
  End-expiratory lung impedance (EELI) detected by using electrical impedance tomography (EIT) 2 minutes after the end of anaesthesia, before the transport in PACU.
End-expiratory lung impedance (EELI) before discharge of PACU. | 5 hours
  End-expiratory lung impedance (EELI) detected by using electrical impedance tomography (EIT) before the discharge from PACU (two hours after admission to PACU).
Changes in silent spaces after the end of induction before the surgical procedure. | 1 hour
  Proportion of poorly ventilated lung areas (silent spaces) detected by using after the end of induction before the surgical procedure.
Changes in silent spaces after the end of anaesthesia. | 3 hours
  Proportion of poorly ventilated lung areas (silent spaces) detected by using electrical impedance tomography (EIT) 2 minutes after the end of anaesthesia, before the transport in PACU.
Changes in silent spaces at the end of the surgical procedure. | 3 hours
  Proportion of poorly ventilated lung areas (silent spaces) detected by using electrical impedance tomography (EIT) at the end of the surgical procedure.
Changes in silent spaces before discharge of PACU. | 5 hours
  Proportion of poorly ventilated lung areas (silent spaces) detected by using electrical impedance tomography (EIT) before the discharge from PACU (two hours after admission to PACU).
Ventilation inhomogeneity after the end of anaesthesia. | 3 hours
  Ventilation inhomogeneity detected by using electrical impedance tomography (EIT) 2 minutes after the end of anaesthesia, before the transport in PACU.
Ventilation inhomogeneity before discharge of PACU. | 5 hours
  Ventilation inhomogeneity detected by using electrical impedance tomography (EIT) before the discharge from PACU (two hours after admission to PACU).
Ventilation inhomogeneity after the end of induction before the surgical procedure. | 1 hour
  Ventilation inhomogeneity detected by using electrical impedance tomography (EIT) after the end of induction before the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fuchs, PD MD, Principal Investigator — University of Bern
Locations (2):
- Switzerland (2):
  - Inselspital, Bern
  - University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: No